CLINICAL TRIAL: NCT07374822
Title: Study on the Real-World Eradication Success Rate of Helicobacter Pylori Infection and Its Influencing Factors
Brief Title: Real-World Study of Helicobacter Pylori Eradication Success and Its Determinants
Status: Completed | Type: Observational
Sponsor: Run-hua Li (Other)
Responsible Party: Sponsor-Investigator, Run-hua Li, Clinical Physician and Principal Research Investigator, Shenzhen Hospital of Southern Medical University
Organization: Shenzhen Hospital of Southern Medical University (Other)
Other Study IDs: NYSZYYEC2024K049R002
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2024-05

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori; H. pylori eradication; Real-world study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Helicobacter pylori Infection: Participants who underwent H. pylori testing and/or eradication treatment at Shenzhen Hospital of Southern Medical University between 2016 and 2023.
  This cohort includes patients receiving different eradication regimens as part of routine clinical care. No study-assigned interventions are provided.
  Interventions: Other: No Study-Assigned Intervention

INTERVENTIONS:
Other: No Study-Assigned Intervention — Participants receive standard-of-care H. pylori eradication regimens as determined by their treating physicians.
  The study does not assign or modify any treatment. Data are collected retrospectively from routine clinical records.

SUMMARY:
This study aims to evaluate the real-world effectiveness of different treatment regimens used to eradicate Helicobacter pylori (H. pylori) infection in routine clinical practice. H. pylori is a common bacterial infection that can lead to chronic gastritis, peptic ulcers, and gastric cancer. Treatment success varies widely in real-world settings due to factors such as antibiotic resistance, patient characteristics, and treatment adherence.

This retrospective observational study will review medical records of patients who underwent H. pylori testing and/or eradication treatment at Shenzhen Hospital of Southern Medical University between 2016 and 2023. No additional tests, visits, or interventions will be performed beyond standard clinical care. The study will collect information on demographics, comorbidities, treatment regimens, test results, and eradication outcomes.

The primary goal is to determine the real-world eradication success rate of commonly used treatment regimens. A secondary goal is to identify factors that may influence treatment effectiveness. Findings from this study may help clinicians choose more effective treatment strategies and improve patient outcomes in everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 14 years.
* Patients who underwent Helicobacter pylori (H. pylori) testing and/or eradication treatment at Shenzhen Hospital of Southern Medical University between 2016 and 2023.
* Diagnosis of H. pylori infection based on the Sixth National Consensus Report on the Management of Helicobacter pylori Infection (Non-Eradication Section) or clinically accepted testing methods.

Exclusion Criteria:

* Children younger than 14 years old.
* Pregnant or breastfeeding women.
* Patients deemed unsuitable for participation by the investigator based on clinical judgment.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients who underwent Helicobacter pylori (H. pylori) testing and/or eradication treatment at Shenzhen Hospital of Southern Medical University between 2016 and 2023. These patients represent a real-world clinical population receiving routine diagnostic evaluation and standard-of-care treatment for H. pylori infection. Individuals aged 14 years and older, regardless of sex, are eligible for inclusion. Patients may present with various gastrointestinal or systemic comorbidities commonly associated with H. pylori infection. No study-specific interventions are administered, and all treatments are determined by the patients' treating physicians as part of usual clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
H. pylori Eradication Success Rate | Within 4-12 weeks after completion of eradication therapy
  The proportion of patients who achieve successful eradication of Helicobacter pylori, as confirmed by a urea breath test (C13), stool antigen test, histology, or other clinically accepted diagnostic methods.
  Eradication success is defined as a negative post-treatment test result.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] https://rs.yiigle.com/cmaid/1435828

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT07374822/Prot_SAP_000.pdf